CLINICAL TRIAL: NCT06509919
Title: Application of a Model Based on Plasma cfDNA Fragmentomics in the Early Diagnosis of Prostate Cancer.
Brief Title: Application of a Novel Biomarker Based on Plasma cfDNA Assay in the Early Diagnosis of Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Ningbo No. 1 Hospital (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Jiangsu Provincial People's Hospital (Other); The First Affiliated Hospital of Soochow University (Other); West China Hospital (Other); Zhongda Hospital (Other); Northern Jiangsu People's Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ren Shancheng, Professor，Chief of Urology, Shanghai Changzheng Hospital
Other Study IDs: KAL1
Record Dates: First submitted 2024-07-14; First posted 2024-07-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: Elevated PSA; Biopsy; Prostate cancer; Prostate neoplasms; cfDNA; Machine learning
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with elevated PSA test results (4-10ng/ml)
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — Before undergoing a prostate biopsy, participants will have about 10 mLs of venous blood drawn. Blood will be sent to Geneseeq Technology Inc. for whole genome high-throughput sequencing of plasma cfDNA.

SUMMARY:
The goal of this diagnostic test is to obtain multiple cell-free DNA （cfDNA） fragment profiles of subjects by whole genome sequencing based on plasma cfDNA, build a prostate cancer prediction model by machine learning, and to validate the efficacy of this model in patients who need to undergo needle prostate biopsy base on their prostate-specific antigen（PSA） or clinical or imaging evidence. Therefore, this study aims to explore the efficacy of this prostate cancer prediction model in distinguishing between patients with PSA "gray zone" (4-10 ng/ml) in the diagnosis of prostate cancer and patients with clinically significant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male, 18-80 years old;
2. PSA: 4-10ng/ml;
3. Patients scheduled for prostate biopsy：

   * fPSA（free PSA）/PSA < 0.16 or PSAD（PSA density） > 0.15 (ng/mL/cm³) or PSAV（PSA velocity） > 0.75 (ng/mL/year) ② positive DRE （digital rectal examination） ③suspicious positive lesions on ultrasound/MRI).

Exclusion Criteria:

1. Patients with a prior diagnosis of any malignancy within 5 years;
2. Patients who have undergone prior transurethral resection or enucleation of the prostate;
3. Patients who have received prior treatment for prostate cancer, including but not limited to endocrine therapy, targeted therapy, and immunotherapy;
4. Patients with long-term use of anticoagulant and antiplatelet aggregation drugs (anticoagulant discontinued for less than 1 week);
5. Received any form of oncological treatment, including surgery, radiotherapy/chemotherapy, endocrine therapy, targeted therapy, and immunotherapy prior to enrollment for blood sampling;
6. concurrently suffering from other serious systemic diseases that, in the opinion of the investigator, may interfere with the treatment, evaluation and compliance of this trial, including serious respiratory, circulatory, neurological, psychiatric, gastrointestinal, endocrine, immune, urinary and other systemic diseases;
7. Organ transplant recipients or prior non-autologous (allogeneic) bone marrow or stem cell transplant population;
8. Subjects who have had a blood transfusion 1 month prior to the blood draw;
9. Patients who are participating in other clinical trials, or who have participated in other clinical trials that have been completed less than 1 year ago;
10. Patients who, in the judgment of the investigator, are not suitable for participation in this clinical trial;
11. Patients who meet any of the above criteria may not be included as subjects.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients aged 18-80 with PSA tests score of 4-10 ng/ml and are scheduled for a prostate biopsy.
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-07-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
AUROC value for predicting positive needle biopsy results (prostate cancer) in individuals with PSA levels in the gray zone. | Through completion of study and all data analysis which may take up to one and a half years.
Sensitivity for predicting positive needle biopsy results (prostate cancer) in individuals with PSA levels in the gray zone. | Through completion of study and all data analysis which may take up to one and a half years.
Specificity for predicting positive needle biopsy results (prostate cancer) in individuals with PSA levels in the gray zone. | Through completion of study and all data analysis which may take up to one and a half years.

SECONDARY OUTCOMES:
AUROC value for predicting clinically significant prostate cancer (GS > 7) in pathological results. | Through completion of study and all data analysis which may take up to one and a half years.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzheng hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No